CLINICAL TRIAL: NCT07264296
Title: Implant-related Infections in Patients With Skeletal Sarcomas
Acronym: IRISSAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other); The Swedish Society of Medicine (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-04459-01; Dnr 2023-04459-01 (Other: Etikprövningsmyndigheten); 2022-00853 (Other Grant/Funding Number: Swedish Research Council); ALFGBG-978896 (Other Grant/Funding Number: The ALF agreement); GLS-973592 (Other Grant/Funding Number: The Gothenburg Society of Medicine); LU2021-0048 (Other Grant/Funding Number: IngaBritt and Arne Lundberg Foundation)
Record Dates: First submitted 2025-05-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Implant Infection; Skeletal Sarcoma; Hip Arthritis; Prosthesis-Related Infections; Knee Arthritis
Keywords: Biofilm; Periprosthetic joint infection; Skeletal sarcoma
MeSH Terms: conditions — Osteosarcoma; Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone, blood, joint fluid and tissue samples will be obtained. In the case of infection, bacterial strains will be retained in a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Skeletal sarcoma group: Patients who receive a megaprosthesis as a primary procedure for skeletal sarcoma.
- Periprosthetic joint infection after skeletal sarcoma: Patients with a periprosthetic joint infection after surgery with a megaprosthesis due to skeletal sarcoma.
- Periprosthetic joint infection after hip/knee replacement due to osteoarthritis: Non-immuncompromised patients with periprosthetic joint infection following a primary total hip or knee replacement.

SUMMARY:
The aim of this observational study is to gain knowledge on the microbial and immunological factors behind implant-related infections in patients with skeletal sarcoma.

The main research question the project aims to answer is:

• Are immunological factors more important than microbial factors in peri-prosthetic joint infections in orthopaedic oncology patients?

Patients with skeletal sarcoma planned for primary surgery (tumour resection and replacement with a megaprosthesis) will be sampled intraoperatively to obtain a cross-section bone tissue slice at the resection margin, three soft tissue biopsies and joint fluid (if possible). Patients who develop a peri-prosthetic joint infection after their primary surgery will be sampled in a similar manner during revision surgery.

An additional group of patients with periprosthetic joint infection of a hip or knee prosthesis due to osteoarthritis will be sampled during their revision surgery (bone biopsies, soft tissue biopsies and joint fluid, if possible).

Blood samples will be taken from all patients pre-operatively for extensive biochemical and cellular analyses.

Researchers will compare periprosthetic tissues before and after infection. Further, periprosthetic infected tissues in patients treated for skeletal sarcoma will be compared to periprosthetic infected tissues in patientens treated for osteoarthritis. This will be done to attempt to identify host and microbial mechanisms responsible for the increased infection rate in patients with a megaprosthesis due to skeletal sarcoma (infection incidence rate up to 30%) compared to patients with a hip or knee prosthesis due to osteoarthritis (infection incidence rate 1-2%).

DETAILED DESCRIPTION:
In orthopaedic oncology, the risk and consequences of orthopaedic device related infections (ODRIs) are heightened as the patients often have compromised immune responses due to underlying disease, chemotherapy or radiation. The implants used may be weight-bearing to the extent that they are impossible to remove or exchange in case of infection, and thereby, in worst case, resulting in amputation or death. Compared to the 1-2% incidence of PJI in a non-oncological population with a total hip- or knee prosthesis, patients with a megaprosthesis due to skeletal sarcoma have an infection incidence of 3-25%. Patient-related factors, extensive and repeated surgery and large reconstructive implants likely account for the increased incidence.

To our knowledge no study has evaluated the role of microbiological factors such as the biofilm production and susceptibility in this population. Further, deficient immunological factors in these patients, such as defect neutrophil migration, cytokine expression and phagocyte respiratory burst, involved in the killing of microbes, may provide an environment favouring more virulent phenotypes. Fundamental knowledge on the role of biofilm in this population could add to the improvement in treatment planning and outcome.

Distinguishing causative pathogens from contaminants may be challenging, especially in polymicrobial infections. The addition of metagenomic diagnostics, still sparsely used in clinical practice, may improve sensitivities, but predictive accuracy is still an issue. Comparing the results of conventional microbiological culturing with metagenomic sequencing would be of interest to determine the accuracy of current diagnostic methods.

The present study is an exploratory project addressing the multifactorial nature of PJI focusing on microbial phenotype in patients with skeletal sarcoma. The role of host, microbe and implant factors will be investigated using a set of different methods and compared to cases och PJI in patients will a conventional hip- or knee prosthesis.

Pre-operative blood samples will be taken and samples of peri-prosthetic soft tissue, bone and joint fluid will be collected intra-operatively. Patients will be sampled during their primary operation with a megaprosthesis due to skeletal sarcoma and in case of postoperative PJI, they will be sampled in the same manner during their revision surgery. Patients undergoing a reoperation due to PJI in a conventional total hip- or knee prosthesis will also be sampled with blood, bone, soft tissue and joint fluid intraoperatively.

Descriptive comparisons between (i) periprosthetic tissues and PJI tissues before and after infection in orthopaedic oncology patients, and (ii) PJI tissues in orthopaedic oncology and conventional PJI patients, will be made in regard to the following parameters:

Role of the host:

* Clinical parameters: ASA-score, diabetes, BMI, age, sex, antibiotic use 2 weeks prior to surgery, duration of chemotherapy, type of chemotherapy, chemotherapy cessation, symptom onset in case of infection, implant type, surgery duration, osteosarcoma type, grade and stage, location of surgery, length of resection.
* Biochemistry in blood (complete white blood cell count with differential, density of neutrophils, CRP, procalcitonin, IL-6).
* Histology and immunohistochemistry (FISH for identification of bacteria, inflammatory infiltrates (presence of foreign body giant cells), angiogenesis, tissue necrosis)
* Gene expression (markers related to angiogenesis, inflammation, microbial recognition and tissue necrosis). In selected paraffin-embedded samples, analysis with spatial transcriptomics will be explored.

Role of the pathogen:

* Five tissue cultures for routine culturing (to determine the causative agent) and one additional for bacterial DNA extraction and 16S rRNA gene sequencing.
* Clinical staphylococcal strains isolated from PJI and tumour endoprosthesis at time of infection will be characterised and compared with respect to their phenotypic biofilm production, antimicrobial susceptibility and presence of virulence genes using CV, MBEC and NGS.
* Difference in gene expression of biofilm-related genes between staphylococcal PJI strains (conventional & orthopaedic oncology) when grown on titanium with serum pre-conditioning in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with skeletal sarcoma planned for primary surgery with resection of tumour and replacement with a megaprosthesis.
* Patients operated with a megaprosthesis due to skeletal sarcoma who develop a peri-prosthetic joint infection (PJI).
* Patients diagnosed with PJI after total hip or knee replacement due to osteoarthritis.

Exclusion Criteria:

* None in the group of patients with skeletal sarcoma.
* Patients in the PJI group who have a total hip or knee replacement are excluded if they use immunomodulary medication or have a immunodeficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of patients will be studied:
  * Patients who undergo surgery with a megaprosthesis due to skeletal sarcoma
  * Patients who have a PJI of a megaprosthesis
  * Patients who have a PJI after total hip or knee replacement due to osteoarthritis
  All patients will be recruited consecutively at the Sahlgrenska University Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in virulence properties in causative microbes in the two groups of PJI | Sampling will occur intraoperatively, bacteria will be frozen, no time frame neccessary
  A descriptive analysis of genotype will be conducted

SECONDARY OUTCOMES:
Differences in periprosthetic tissues in the two PJI groups | Sampling will occur intraoperatively, tissues will be preserved, no time frame neccessary
  Descriptive analysis of periprosthetic tissue using histological methods

OTHER OUTCOMES:
Differences in biofilm production ability between causative microbes in the two PJI groups | Sampling will occur intraoperatively, bacteria will be frozen, no time frame neccessary
  Biofilm production will be assesed and categorised into none/weak and moderate/strong

CONTACTS AND LOCATIONS:
Overall Officials: Karin Svensson Malchau, PhD, Principal Investigator — Vastra Gotaland Region; Margarita Trobos, Assoc Prof, Principal Investigator — Göteborg University
Locations (1):
- Ortopedi, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
The main results will be presented at an aggregated level. In some cases, individual data may be presented (e.g. characteristics of a bacterial strain in relation to clinical outcome), but this information will be unidentified so that it cannot be deduced to the individual.
  All compiled personal data will be stored on a password-protected hospital server that only the research group has access to. No personal data will be reported in publications.
  The results of the study will be documented according to the study protocol and placed in a journal. Participants will be coded in a document together with the social security numbers.
  Information about the participants, their health and the code key will be collected at the Orthopaedic Clinic where it will be treated confidentially and securely for 10 years. The handling of the participants' information is regulated by the Personal Data Act (SFS 1998: 204).